CLINICAL TRIAL: NCT00868062
Title: Do 100 kiloDaltons Matter? A Prospective Randomised Double-blind Study on the Blood Volume Expanding Effects of Two Different Colloids in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Responses to Colloid Infusions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Sherwood Forest Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 08101 colloidAug08
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: The responses of patients to 1L infusions of Gelofusine (succinylated gelatine 40g/L) and Voluven (6% hydroxyethyl starch in 0.9% saline) intraoperatively.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Succinylated gelatine, 40g/L, (Gelofusine - B Braun)

INTERVENTIONS:
Other: Succinylated gelatine, 40g/L, (Gelofusine - B Braun) — 1 litre infusion following induction of anaesthesia

SUMMARY:
In situations such as dehydration, illness and surgery, fluid 'drips' are given to patients to keep them hydrated. Different fluids stay in the circulation for different lengths of time. For example, some types of fluid remain in the circulation for a short time which means patients would need to be given more fluid to achieve the desired effects. Giving a lot of fluid to sick patients can in itself cause problems, for example, it can affect the way the bowels work and delay the patient's recovery from illness. In these situations the investigators use specialized fluids called colloids, that are designed to stay in the circulation for longer. This means a smaller amount of fluid needs to be used and less problems are likely to occur. There are two different types of colloids that are commonly used, but the investigators do not know which of them is better. The purpose of this study is to investigate which of the two different colloids (one is called Gelofusin and the other is called Voluven) works better in patients who undergo surgery. Knowing which of the two fluids works best in patients will help us improve the care of surgical patients. The investigators hypothesis is that the fluid that has the larger size of molecules as part of the solution will work better during surgery.

DETAILED DESCRIPTION:
To study the responses of patients to 1 litre infusions of Gelofusine (succinylated gelatine 40g/L) and Voluven (6% hydroxyethyl starch in 0.9% saline) over 1 h intraoperatively. In particular, the extent and time course of the effects of the two infusions on haematocrit, serum albumin, serum biochemistry, plasma expanding capacity and the resultant urinary responses will be measured

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-60 years undergoing elective laparoscopic cholecystectomy for proven gallstone disease.
* BMI of 20-26 kg/m2
* Able to give voluntary written informed consent to participate in the study
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures
* (Females of child bearing age will be offered a pregnancy test)

Exclusion Criteria:

* Patients with a known history of allergic reaction to the colloid infusions
* Patients with acute cholecystitis or the systemic inflammatory response syndrome
* Patients with a serum bilirubin > 25 μmol/l
* Females who are pregnant or refuse to have a pregnancy test
* Patients with a haemoglobin < 10 g/l
* Patients with a history of acute pancreatitis
* Patients likely to undergo common bile duct exploration
* Patients with renal impairment, ischaemic heart disease, cardiac failure and chronic restrictive airways disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The magnitude and duration of the plasma volume expanding effects of the two colloids. | 4 hours

SECONDARY OUTCOMES:
To determine the effects of the two infusions on serum and urinary osmolality, sodium, potassium, chloride, bicarbonate, urea, albumin, microalbumin and haematological parameters. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Lobo, FRCS, Principal Investigator — University of Nottingham; Mukul Dube, FRCS, Principal Investigator — Sherwood Forrest Hospitals NHS Trust
Locations (1):
- Sherwood Forest Hospitals NHS Foundation Trust, Mansfield, Nottinghamshire, United Kingdom